CLINICAL TRIAL: NCT05329337
Title: Seeking a Link Between the Capacity of Peripheral Mononuclear Cells to Induce Insulin Resistance and the Development of Hyperinsulinemia in a General Population
Brief Title: Link Between the Peripheral Mononuclear Cells' Capacity to Induce Insulin Resistance and Hyperinsulinemia
Acronym: IRACTIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Caisse Primaire d'Assurance Maladie du Gard (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: NIMAO/2020-1/PC-01; 2021-A03189- 32 (Other: EudraCT)
Record Dates: First submitted 2022-04-06; First posted 2022-04-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Insulin Resistance; Hyperinsulinism; Immune System
Keywords: Insulin resistance
MeSH Terms: conditions — Insulin Resistance; Hyperinsulinism | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: This is a two-center proof-of-concept study, ancillary to the MetACTIV study, whose objective is to define immune activation profiles from the data of individuals followed by the Gard health insurance fund. The IRACTIV study will include a subset of volunteers from the MetACTIV study for whom a blood sample will be taken as part of the IRACTIV study.
  In order to study the evolution of insulin levels in volunteers, we need to be able to ensure a longitudinal analysis, which requires a link with the MetACTIV study data for the volunteers included in the IRACTIV study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 patients with high insulin levels (13.3 ± 9.2 microU/mL) and markers of metabolic syndrome (Experimental): These are individuals who were isolated from the previous MetACTIV study due to their specific immune profile (Profile 2) defined by 43 immune activation markers and characterized by a high percentage of differentiated T cells and activated T cells.
  Interventions: Diagnostic Test: Blood test
- 20 patients with other immune profiles (Active Comparator)
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Sixteen mL of blood will be collected on EDTA for the purpose of this study

SUMMARY:
This is a two-center proof-of-concept study, ancillary to the MetACTIV study, whose objective is to define immune activation profiles from the data of individuals followed by the Caisse Primaire d'Assurance Maladie du Gard (health insurance fund).

The IRACTIV study will include a subset of volunteers from the MetACTIV study for whom a blood sample will be taken as part of the IRACTIV study.

DETAILED DESCRIPTION:
The local health insurance fund regularly offers people who have already had a free health check-up the opportunity to re-do a check-up. This invitation will be made as part of the routine, by mail. People who have participated in the MetACTIV study will be asked to participate in the present IRACTIV study ( they will be sent an information note). That way, up to 30 volunteers who previously participated in the MetACTIV study, including 10 for whom a particular profile has been identified will be recruited again in sequence.

On the day of consultation at the Gard health insurance fund, consent will be collected from subjects who have agreed to participate. The participation of the volunteers will be reduced to this single visit and 16 mL of blood will be collected on EDTA for the purpose of this study. As in the previous MetACTIV study, this blood will be transported to the Biological Resource Center at Nîmes University Hospital. From this blood, the plasma will be frozen and stored at -80°C for subsequent determination of insulin levels under the same conditions as for the MetACTIV study. Peripheral blood mononuclear cells will be frozen and, later, cultured at the Institute of Human Genetics in complete medium for 48 hours. The effect of the supernatants of these cultures on Akt phosphorylation in HepG2 cells exposed to 10nM of insulin will then be quantified by two different techniques (Western Blot and ELISA). This effect will be expressed as a percentage of inhibition compared to the phosphorylation of Akt induced by insulin alone. The insulin slope between the measurement performed in the MetACTIV study and this IRACTIV study will also be calculated and compared to the peripheral blood mononuclear cells ability to induce insulin resistance in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who participated in the MetACTIV study.
* Profile 2 subgroup-specific inclusion criteria:
* MetACTIV study individual with a Profile 2.
* Persons who have given free informed consent.
* Persons who have signed the consent form.
* Persons affiliated to or benefiting from a health insurance plan.
* Adults (≥18 years of age).

Exclusion Criteria:

* Persons participating in Category 1 research involving human subjects
* Persons in an exclusion period as determined by another study.
* Persons under court protection, guardianship or trusteeship.
* Persons who are incapable of giving consent.
* Persons for whom it is impossible to give clear information.
* Pregnant, parturient or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose | Day 0
  Fasting blood glucose will be measured during a routine health evaluation and measured in mM/L.
End-of-study insulinemia | Month 18
  The amount of insulin in the blood of patients will be measured during a routine health evaluation and measured in µU/L.
Effect of peripheral blood mononuclear cell supernatant on intensity of the signal induced by insulin in hepatocytes. | Hour 48
  Peripheral blood mononuclear cells are isolated on a Ficoll gradient and frozen. These frozen peripheral blood mononuclear cells will be sent to the Institute of Human Genetics for culture and supernatants will be recovered after 48 hours. The effect of these supernatants on insulin signaling will then be tested. To do so, they will be added or not to cultured HepG2 cells stimulated 24 hours later by 10nM insulin. After stimulation, HepG2 cells will be lysed and their total Akt and phosphorylated Akt content measured by ELISA and Western Blot. The proportion of phosphorylated Akt in HepG2 cells exposed to peripheral blood mononuclear cells supernatant will be compared with the proportion of phosphorylated Akt in HepG2 cells not exposed to peripheral blood mononuclear cells supernatant and expressed as the percentage of insulin signaling inhibition induced by the peripheral blood mononuclear cells supernatant.

SECONDARY OUTCOMES:
A. Percentage inhibition of Akt phosphorylation in Profile 2 patients compared with other immune profiles. | Hour 48
  The decrease in signal intensity induced in hepatocytes by insulin induced by peripheral blood mononuclear cell supernatant from volunteers with Profile 2 will be compared to the decrease in this intensity induced by peripheral blood mononuclear cell supernatant from volunteers with another immune activation Profile. Measured as a percentage.
B. Increase in insulinemia over time in Profile 2 patients compared with other immune profiles. | Month 18
  Insulinemia in Profile 2 volunteers, measured in µU/mL, will be compared with that of other immune profiles.

OTHER OUTCOMES:
Age of Profile 2 patients | Day 0
  In years
Weight of profile 2 patients | Day 0
  In kg
Gender of Profile 2 patients | Day 0
  male / female
Waist measurement of Profile 2 patients | Day 0
  In cm
Hip circumference of Profile 2 patients | Day 0
  In cm
Systolic blood pressure in Profile 2 patients | Day 0
  In mmHg
Diastolic blood pressure in Profile 2 patients | Day 0
  In mmHg
High-density lipoproteins in Profile 2 patients | Day 0
  mM/L
Low-density lipoproteins in Profile 2 patients | Day 0
  mM/L
Triglycerides in Profile 2 patients | Day 0
  mM/L
Hemoglobin A1c in Profile 2 patients | Day 0
  mM/L

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire, Nîmes, Gard
  - Caisse Primaire d'Assurance Maladie du Gard, Nîmes, Gard

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kundura L, Cezar R, Ballongue E, Andre S, Michel M, Mettling C, Lozano C, Vincent T, Muller L, Lefrant JY, Roger C, Claret PG, Duvnjak S, Loubet P, Sotto A, Tran TA, Estaquier J, Corbeau P. Low Percentage of Perforin-Expressing NK Cells during Severe SARS-CoV-2 Infection: Consumption Rather than Primary Deficiency. J Immunol. 2024 Apr 1;212(7):1105-1112. doi: 10.4049/jimmunol.2300359. PMID 38345346